CLINICAL TRIAL: NCT03978312
Title: Implications of Nutrition Health Literacy on Accessibility and Engagement With Nutrition Information in Cancer Patients and Their Support Networks
Brief Title: Nutrition Health Literacy of Cancer Patients and Their Support Networks.
Acronym: NiiCproject
Status: Terminated | Type: Observational
Why Stopped: Recruitment was due to be extended (March 20) due to slow initial recruitment however was terminated early due to corresponding arrival of COVID-19 to UK. (16 recruited to cultural and linguistic phase and 42 to observational cohort)
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Macmillan Cancer Support (Other); University of Kansas (Other); Bishop Grosseteste University (Unknown); Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 18ON105
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Oncologic Disorders; Haematological Malignancy; Nutrition Aspect of Cancer
Keywords: Nutrition; Health; Literacy; Education; Information; Knowledge
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Literacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nominal consensus group — NLit-UK linguistic and cultural adaptation (NLit-UK) 2 x nominal consensus groups evidence review and topic expert engagement
Other: Observational cohort (validity and reliability testing) — Nutrition Literacy Measurement Tool validation (NLit-UK). Target sample 366 on treatment cancer patients confirmatory binary analysis for validity and reliability.

SUMMARY:
An exploration of the impact of nutrition literacy on ability of cancer patients and their support networks to get, understand and use nutrition information during cancer treatment.

DETAILED DESCRIPTION:
The study is composed of two component projects:

Project A: Validation of a NLit tool for UK population.

NLit tool is a measurement tool developed at Kansas University to measure nutrition health literacy. It assesses the following functional literacy skills: numeracy & literacy and the following nutrition knowledge fields: macronutrients, food labels, portion sizes, food groups and consumer skills.

This project has two phases:

Phase A: Nominal consensus groups x 2 - consumer adaptation and tool review for UK use and pilot testing of electronic tool.

Phase B: Testing adapted tool in a group of cancer patients for statistical validation.

Project B: Planned survey of people with cancer and their families to explore experiences of access to nutrition information

This survey is a combination of validated and unvalidated questions built on models of nutrition health literacy. With validated fields being used to evaluate and understand responses to unvalidated questions.

It explores access to nutrition information, self-efficacy, confidence, health care infrastructure and support with nutrition information, population demographics, food security, sources of nutrition information, perceived practical skills and knowledge base.

ELIGIBILITY:
NLit-UK development

Inclusion Criteria:

* Members of the public (carers, health service users, lay persons)
* Cancer patients with confirmed diagnosis
* Friends or family members supporting a patient with a confirmed diagnosis of cancer
* > 18 yrs old
* Received cancer treatment at Nottingham University Hospitals between Jan 15 and March 20

Exclusion Criteria:

* Paediatrics < 18yrs at the time of diagnosis and treatment
* Unconfirmed diagnosis of cancer
* Patients on watch and wait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Cancer patients
  * Friends or family of cancer patients
  * Members of the public
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Nutrition health literacy - UK | Jun 19 - Mar 2020
  Measured by UK modified NLit developed during study cultural and linguistic modification of (Gibbs et al., 2018 - original validation) - 64 item questionnaire
  Scoring interpretation from study: NLit-UK (63item) and NLit-UK short (42-item) NLit-UK (63-item): Scoring interpretation is ≤44 correct is "likelihood of poor nutrition literacy"; 45-57 is "possibility of poor nutrition literacy"; and scores ≥58 is "likelihood of good nutrition literacy
  NLit-UK short (42-item): Scoring interpretation is ≤28 correct is "likelihood of poor nutrition literacy"; 29-37 is "possibility of poor nutrition literacy"; and scores ≥39 is "likelihood of good nutrition literacy
NVS-UK health literacy | Jun 19 - Mar 2020
  Validated tool - 6 part question (Rowlands et al, 2013)
  Scoring interpretation: low health literacy (≤1), intermediate health literacy (2-3), adequate health literacy (≥4).

SECONDARY OUTCOMES:
Prior Knowledge | Jun 19 - Mar 2020
  Did you receive any nutrition advice as part of your care for any of these conditions?" (Yes or No).
Educational status (modified HINTS4 Cyc1) | Jun 19 - Mar 2020
  What is the highest grade or level of schooling you completed? GCSE D or less/ GCSE C or above/ Unsure
Economic status (modified HINTS 2) | Jun 19 - Mar 2020
  At the end of the month, how much money are you able to put aside? (Nothing, £100 or less, £101-250, £251-500, £501-1000, more than £1000, do not want to say).
How important did you consider nutrition was in helping you through your treatment? | Jun 19 - Mar 2020
  Response sets: Didn't know enough to consider / Not important ; Moderately Important; Very or extremely important

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Miller, MBiol, PgDip, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbs HD, Ellerbeck EF, Befort C, Gajewski B, Kennett AR, Yu Q, Christifano D, Sullivan DK. Measuring Nutrition Literacy in Breast Cancer Patients: Development of a Novel Instrument. J Cancer Educ. 2016 Sep;31(3):493-9. doi: 10.1007/s13187-015-0851-y. PMID 25952941
- [Background] Gibbs HD, Ellerbeck EF, Gajewski B, Zhang C, Sullivan DK. The Nutrition Literacy Assessment Instrument is a Valid and Reliable Measure of Nutrition Literacy in Adults with Chronic Disease. J Nutr Educ Behav. 2018 Mar;50(3):247-257.e1. doi: 10.1016/j.jneb.2017.10.008. Epub 2017 Dec 12. PMID 29246567
- [Background] Gibbs HD, Harvey S, Owens S, Boyle D, Sullivan DK. Engaging Experts and Patients to Refine the Nutrition Literacy Assessment Instrument. BMC Nutr. 2017;3:71. doi: 10.1186/s40795-017-0190-y. Epub 2017 Aug 22. PMID 28890794